CLINICAL TRIAL: NCT06505850
Title: Comparisons of Postoperative Sore Throat and Subglottic Airway Injury Between Endotracheal Tubes with Different Cuff Shapes in Breast Cancer Patients
Brief Title: Cuff Shape and Postoperative Sore Throat in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Wei-Cheng Tseng, Principal Investigator, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: A202405086_V3
Record Dates: First submitted 2024-07-01; First posted 2024-07-17 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer; Postoperative Sore Throat; Subglottic Airway Injury; Endotracheal Tube Cuff
Keywords: Endotracheal tube cuff; Postoperative sore throat; Subglottic airway injury; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Tapered-shaped cuff ETT group (Experimental): A tapered-shaped cuff tube was used to intubate for general anesthesia
  Interventions: Device: Tapered-shaped cuff tracheal tube
- Cylindrical-shaped cuff ETT group (Active Comparator): A cylindrical-shaped cuff tube was used to intubate for general anesthesia
  Interventions: Device: Cylindrical-shaped cuff tracheal tube

INTERVENTIONS:
Device: Tapered-shaped cuff tracheal tube — Tracheal intubation with a tapered-shaped cuff tube
  Arms: Tapered-shaped cuff ETT group
Device: Cylindrical-shaped cuff tracheal tube — Tracheal intubation with a cylindrical-shaped cuff tube
  Arms: Cylindrical-shaped cuff ETT group

SUMMARY:
This study aimed to evaluate the impact of endotracheal tube cuff shapes on the incidence and severity of postoperative sore throat

DETAILED DESCRIPTION:
Postoperative sore throat (POST) is a minor complication after general anesthesia with tracheal intubation but may negatively affect patient satisfaction and postoperative recovery. Due to the multifactorial nature, the detailed mechanism of POST has not been fully understood. However, mucosal irritation and inflammation related to the presence of an ETT within the trachea appear to be one of the primary causes of POST, which may involve elements including the tube size, intracuff pressure, and duration of intubation. In addition, the cuff design of an ETT, which can determine the contact area between the cuff and the tracheal mucosa, is reported to affect the development of POST. This study aimed to evaluate the impact of endotracheal tube (ETT) cuff shapes on the incidence and severity of POST. Additionally, we investigated the influence of ETT cuff shapes on the degree of subglottic injury following GA for breast cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female patients scheduled for elective breast cancer surgery performed in the supine position requiring tracheal intubation

Exclusion Criteria:

* Age < 18 years or age > 80 years
* Diseases or anatomic abnormalities in the neck, larynx, or pharynx
* Combined surgery such as breast reconstruction
* Active pulmonary disease
* Morbid obesity (body mass index ≥ 40 kg/m2)
* Pregnancy
* Refusal to join the study

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients scheduled for elective breast cancer surgery performed in the supine position requiring tracheal intubation
Enrollment: 176 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
The incidence of postoperative sore throat | Postoperative 48 hours
The severity of postoperative sore throat | Postoperative 48 hours
  1, none; 2, mild (complains of sore throat only on asking); 3, moderate (complains of sore throat on her own); 4, severe (change of voice or hoarseness, associated with throat pain)

SECONDARY OUTCOMES:
Intraoperative fentanyl consumption | The end of surgery
Intraoperative propofol consumption | The end of surgery
Intraoperative rocuronium consumption | The end of surgery
The degree of subglottic injury | Intraoperative (The time point at extubation)
  None: no subglottic injury; mild: mucosal hyperemia and edema and/or slight submucosal hematoma; moderate: moderate submucosal hematoma; severe: mucosal laceration and/or mucosal bleeding)

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
There is no plan to share

REFERENCES:
- [Background] Monroe MC, Gravenstein N, Saga-Rumley S. Postoperative sore throat: effect of oropharyngeal airway in orotracheally intubated patients. Anesth Analg. 1990 May;70(5):512-6. doi: 10.1213/00000539-199005000-00008. PMID 2331067
- [Background] Christensen AM, Willemoes-Larsen H, Lundby L, Jakobsen KB. Postoperative throat complaints after tracheal intubation. Br J Anaesth. 1994 Dec;73(6):786-7. doi: 10.1093/bja/73.6.786. PMID 7880666
- [Background] Biro P, Seifert B, Pasch T. Complaints of sore throat after tracheal intubation: a prospective evaluation. Eur J Anaesthesiol. 2005 Apr;22(4):307-11. doi: 10.1017/s0265021505000529. PMID 15892411
- [Background] Lehmann M, Monte K, Barach P, Kindler CH. Postoperative patient complaints: a prospective interview study of 12,276 patients. J Clin Anesth. 2010 Feb;22(1):13-21. doi: 10.1016/j.jclinane.2009.02.015. PMID 20206846
- [Background] El-Boghdadly K, Bailey CR, Wiles MD. Postoperative sore throat: a systematic review. Anaesthesia. 2016 Jun;71(6):706-17. doi: 10.1111/anae.13438. Epub 2016 Mar 28. PMID 27158989
- [Background] Chang JE, Kim H, Han SH, Lee JM, Ji S, Hwang JY. Effect of Endotracheal Tube Cuff Shape on Postoperative Sore Throat After Endotracheal Intubation. Anesth Analg. 2017 Oct;125(4):1240-1245. doi: 10.1213/ANE.0000000000001933. PMID 28368938
- [Derived] Chen GC, Lo KL, Wu ZF, Chan SM, Cheng SY, Ko CL, Chu CM, Tseng WC. Comparison of the incidence and severity of postoperative sore throat and subglottic airway injury with cylindrical versus tapered cuff endotracheal tubes in women undergoing surgery for breast cancer: a randomized controlled trial. BMC Anesthesiol. 2025 Apr 12;25(1):181. doi: 10.1186/s12871-025-03040-y. PMID 40221641